CLINICAL TRIAL: NCT05631600
Title: Manuka Honey as an Adjunct to Non-surgical Periodontal Therapy: Clinical Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Darko Bozic, Associate professor of Periodontology, University of Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-PA-30-IX-9/2019
Record Dates: First submitted 2022-10-26; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontal Bone Loss; Periodontal Attachment Loss
Keywords: Periodontitis; Manuka honey; Periodontal pocket depth
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Alveolar Bone Loss; Periodontal Attachment Loss; Periodontitis

STUDY DESIGN:
Intervention Model Description: Split-mouth study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Manuka honey (Experimental): The intervention in this study was conducted in a split-mouth design, meaning that after completing the NSPT for each subject, Manuka honey was administered as an adjunct to the periodontal treatment in two randomly selected quadrants of the oral cavity around the teeth with a specially designed cannula. The cannula reached the bottom of the periodontal pocket and moved circumferentially around the tooth at 6 sites, and Manuka honey was extruded until the excess of the material was observed in the sulcus.
  Interventions: Biological: Manuka honey

INTERVENTIONS:
Biological: Manuka honey — The honey was applied with special designed cannula. The dosage is not exactly define so we inject the amount of honey until until the excess of the material was observed in the sulcus.

SUMMARY:
The goal of this split-mouth clinical trial is to evaluate the effects of Manuka honey applied into periodontal pockets after initial periodontal therapy (NSPT) in the treatment of stage 3 periodontitis.

The main question it aims to answer is:

• does the adjunct of Manuka honey improve the outcome of the non-surgical periodontal treatment.

The intervention in this study was conducted in a split-mouth design, meaning that after completing the NSPT for each subject, Manuka honey was administered as an adjunct to the periodontal treatment in two randomly selected quadrants of the oral cavity around the teeth with a specially designed cannula.

This was followed by oral hygiene instructions and training. The home-performed oral hygiene procedures were focused on interdental cleaning using dental floss and toothbrushing with regular fluoride-containing toothpaste. The subjects were also instructed not to use any form of oral antiseptic (e.g., chlorhexidine) or antibiotic during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders with good systemic health;
* Non-smokers;
* Presence of at least 20 teeth;
* Untreated moderate to advanced generalized chronic periodontitis according to the 1999 Classification 199 , i.e., generalized stage III periodontitis according to the 2007 Classification

Exclusion Criteria:

* Pregnant and nursing women;
* Antibiotics prescribed for dental or non-dental diseases 6 months before the start of the research;
* Systemic diseases or the use of drugs known to affect periodontal tissues, bleeding parameters;
* Acute oral or periodontal inflammation or infection (pericoronitis, necrotizing periodontal diseases, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket depth | Baseline; 12 months
  Evaluation of changes of periodontal pocket depth
Clinical attachment level | Baseline: 12 months
  Evaluation of changes in terms of clinical attachment gain

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No